CLINICAL TRIAL: NCT03839459
Title: Denosumab for Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Brea Lipe, Associate Professor - Department of Medicine , Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMMY18121
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma; Denosumab
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 120mg of Denosumab will be administered subcutaneously once every 4 weeks

SUMMARY:
This study will assess the safety and tolerability of denosumab in smoldering multiple myeloma subjects as well to see if denosumab can reduce subjects' risk of getting multiple myeloma.

DETAILED DESCRIPTION:
This is an open label, Phase II trial of denosumab 120mg subcutaneous (SC) for patients with smoldering multiple myeloma (SMM). Subjects will be recruited from the James P. Wilmot Cancer Center, University of Rochester in Rochester, New York. Patients seen in the inpatient or outpatient setting with histologically confirmed SMM will be evaluated for this study.

20 patients will be treated as follows: Denosumab: day 1 = 120mg SC every 4 weeks for 12 cycles. Cycles will be 28 days in length. Patients will be followed after completion of the study per standard of care for progression free survival for an additional 2 years after the last dose of denosumab. All patients will take daily vitamin D and calcium supplements of at least 1200mg elemental calcium and 800IU of vitamin D unless documented hypercalcemia develops on study. Pre-existing hypocalcemia must be corrected prior to initiating therapy with denosumab. Serum vitamin D levels will be checked during screening and should be repleted to a total 25-hydroxyvitamin D level ≥30ng/mL.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has confirmed SMM according to the definition of the International Myeloma Working Group (IMWG) definition: serum M-protein ≥3 g/dL or BMPC >10% but less than 60%, or both, along with normal organ and marrow function (CRAB) within 4 weeks prior to baseline. C: Absence of hypercalcemia, evidenced by a calcium ≤11 mg/dL. R: Absence of renal failure, evidenced by a creatinine ≤ 2.0mg/dL A: Absence of anemia, evidenced by a hemoglobin ≥10 g/dL.

   B: Absence of lytic bone lesions per IMWG recommendations:

   One of either PET-CT, low-dose whole-body CT (LDWBCT) or MRI of the whole body or spine. Increased uptake on PET-CT alone is not adequate for the diagnosis of multiple myeloma; evidence of underlying osteolytic bone destruction is needed on the CT portion of the examination.
2. One of the risk factors below that portends for an increased risk of progression to MM:

   * An abnormal free light chain ratio
   * M-spike ≥ 4 g/dL
   * ≥ 50% bone marrow plasma cells
   * Immunoparesis ≥ 20% less than the institutional normal standard of the uninvolved immunoglobulins
3. Serum calcium or albumin-adjusted serum calcium ≥ 2.1 mmol/L (8.4 mg/dL) and ≤ 2.9mmol/L (11.5 mg/dL) (Reference range 8.5-10.8 mg/dL)
4. Able to tolerate daily supplementation of calcium and vitamin D
5. Must have a vitamin D level ≥ 30 ng/mL after repletion
6. Participants must have normal organ as defined below:

   * Total bilirubin ≤ 2.0 x institutional upper limit of normal (ULN); patients diagnosed with Gilbert's syndrome can enroll with a total bilirubin > 2 after review of the principal investigator
   * AST(SGOT) ≤2.5 × institutional ULN
   * ALT(SGPT) ≤2.5 × institutional ULN
7. Age ≥ 18 years.
8. ECOG PS ≤1
9. Life expectancy greater than 12 months
10. Subjects with reproductive potential must be willing to use, in combination with his/her partner, 2 highly effective methods of effective contraception or practice sexual abstinence throughout the study and continue for 5 months after the study duration. Subjects who are surgically sterile (e.g. history of bilateral tubal ligation, hysterectomy) or whose sexual partner is sterile (e.g. history of vasectomy) are not required to use additional contraceptive measures.
11. Ability to understand and the willingness to sign a written informed consent document.

    -Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. Statement on Inclusion of Women and Minorities - Men and women of all ethnicities and racial backgrounds are eligible for this study.

Exclusion Criteria:

1. Prior administration of denosumab.
2. Any history of IV bisphosphonate use prior to or during the study
3. Prescription oral fluorides or bisphosphonate usage > 3 months within the past 2 years
4. Systemic corticosteroids > 10mg prednisone per day
5. Known secondary cause for osteopenia or osteoporosis
6. Patient has symptomatic MM, as defined by any of the following:

   * Lytic lesions or pathologic fractures.
   * Anemia (hemoglobin <10 g/dL)
   * Hypercalcemia (corrected serum calcium > 11.0 mg/dL)
   * Renal insufficiency (creatinine > 2.0 mg/dL).
   * Clonal bone marrow plasma cells > 60%
   * An involved serum free light chain (kappa or Lambda) > 100mg/L with the ratio of the involved/uninvolved free light chains also > 100 mg/L
   * One or more osteolytic lesions on radiography, but more than one lesion is required if < 10% marrow plasma cells. From MRI imaging, there must be more than one lesion of > 5mm in size.
7. Other: symptomatic hyperviscosity, amyloidosis, plasma cell leukemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein)
8. Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw.
9. Active dental or jaw condition that requires oral surgery, including tooth extraction.
10. Non-healed dental/oral surgery, including tooth extraction.
11. Planned invasive dental procedures during the course of study.
12. Evidence of any of the following conditions per subject self-report or medical chart review:

    * Any prior invasive malignancy within 3 years of enrollment that may affect outcome of study
    * Any non-invasive malignancy not treated with curative intent or with known active disease within 3 years before enrollment that may affect outcome of study
    * Major surgery or significant traumatic injury occurring within 4 weeks before enrollment
    * Active infection with Hepatitis B virus or Hepatitis C virus
    * Known infection with human immunodeficiency virus (HIV) requiring IV anti-infective therapy
13. Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment.
14. Female subject of child-bearing potential is not willing to use, in combination with her partner, 2 methods of highly effective contraception during treatment and for 5 months after the end of treatment.
15. Clinically significant hypersensitivity to denosumab or any components of denosumab 120mg.
16. Known sensitivity to any of the products to be administered during the study (e.g., calcium, or vitamin D).
17. Subject is receiving or is less than 14 days since ending other experimental drug (no marketing authorization for any indication).
18. Any major medical or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brea Lipe, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab
Started | 20
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — progression of disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 1
  40-49 | 1
  60-69 | 6
  70-79 | 9
  80-89 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Downgraded Risk of Progression of Smoldering Multiple Myeloma if the Risk Category Decreases.
Description: Risk Categories:
  Low Risk:Patient has SMM, but none of the listed risk factors Low-Intermediate Risk: 1 risk factor is present High-Intermediate Risk: 2 risk factors are present High Risk: 3 risk factors are present
  Risk Factors:
  1. BM plasma cell % ≥50
  2. M-protein ≥ 3g/dL
  3. Involved/ un-involved free light chains ≥ 8
Time Frame: 1 year
Measure: Number; unit: proportion of participants
Arm/Group | Denosumab
Number analyzed (Participants) | 15
proportion of participants | 0

2. Secondary Outcome: Proportion of Subjects With Skeletal Related Events
Description: To be determined by the investigator
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Subjects With Disease Progression to Multiple Myeloma
Description: as for outcome 1
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Subjects With Progression Free Survival
Description: time to progression or death from any cause, whichever occurs first.
Time Frame: 3 year
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Subjects With Change in Bone Mineral Density
Description: baseline and each post-treatment point
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=20)
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Investigations) | 2
Lung infection (Infections and infestations) | 1
Somnolence (Nervous system disorders) | 1
urinary tract infection (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Amnesia (Nervous system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Infections and infestations) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 5
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 6
Endocrine disorders - Other (Endocrine disorders) | 3
Fall (Injury, poisoning and procedural complications) | 4
Fatigue (General disorders) | 12
Fever (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4
General disorders and administration site conditions - Other (General disorders) | 4
Hemoglobin increased (Investigations) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Hypotension (Vascular disorders) | 1
Infections and infestations - Other (Infections and infestations) | 2
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 3
Insomnia (Psychiatric disorders) | 1
Investigations - Other (Investigations) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 9
Malaise (General disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nail infection (Infections and infestations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Nervous system disorders - Other (Nervous system disorders) | 4
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Otitis externa (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Paresthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pharyngitis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 2
Presyncope (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03839459/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03839459/ICF_001.pdf